CLINICAL TRIAL: NCT02653560
Title: Value of Liquid Potassium Magnesium Citrate in Controlling Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU 072012-001
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Potassium; Magnesium; Citrate; DASH
MeSH Terms: conditions — Hypertension | interventions — potassium-magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Potassium magnesium Citrate (KMgCit) arm (Experimental): Potassium magnesium citrate will be prepared by mixing potassium citrate, magnesium citrate and/or citric acid by Meta Pharm Development. The content of each sachet will be dissolved in 250 ml water and will be drunk with breakfast and again with dinner during the KMgCit Phase, to deliver 40 meq K, 20 meq Mg and 74 meq citrate per day for 4 weeks
  Interventions: Drug: Potassium magnesium Citrate (KMgCit)
- Potassium citrate arm (Experimental): A special sachet formulation containing 20 meq K/sachet will be made for the study by Meta Pharm Development. The contents of a sachet will be added to 250 ml water and drunk with breakfast and dinner, to deliver 40 meq K (as citrate) per day during the Potassium Citrate Phase for 4 weeks.
  Interventions: Drug: Potassium citrate powder
- Potassium chloride arm (Experimental): Potassium chloride will contain 20 meq KCl per sachet. During the Potassium Chloride Phase, subjects will dissolve the content of each sachet in 250 ml water and ingest it with breakfast and again with dinner, to deliver 40 meq K (as chloride) per day for 4 weeks
  Interventions: Drug: Potassium chloride powder
- Placebo (Placebo Comparator): Placebo will comprise microcrystalline cellulose, equivalent in volume in each sachet as other test products. During the Placebo Phase, subjects will dissolve the entire content of a sachet in 250 ml water and drink it with breakfast and again with dinner for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Potassium chloride powder
  Arms: Potassium chloride arm
Drug: Potassium magnesium Citrate (KMgCit)
  Arms: Potassium magnesium Citrate (KMgCit) arm
Drug: Potassium citrate powder
  Other Names: Urocit®-K powder
  Arms: Potassium citrate arm
Drug: Placebo
  Arms: Placebo

SUMMARY:
In the DASH (Dietary Approaches to Stop Hypertension) trials, a diet rich in fruits, vegetables, nuts and dairy products, and limited in fat content, was shown to be useful in controlling hypertension. Key components of such a diet are potassium, magnesium and alkali, each of which has been implicated in lowering blood pressure. Whether a liquid formulation of potassium-magnesium citrate will result in equivalent BP effect as the DASH diet is unknown.

DETAILED DESCRIPTION:
The DASH diet is rich in potassium and magnesium. It is also high in alkali content, since the anions are provided mostly by citrate rather than chloride. Considerable data are already available in the literature invoking a protective role on hypertension of potassium, magnesium and alkali.

In this protocol, the investigators want to test the hypothesis that liquid potassium-magnesium citrate (KMgCit) as a pharmaceutical formulation could serve as a surrogate for the DASH diet, and would lower blood pressure among patients with pre- or Stage I hypertension on their customary diet.

Each subject will participate in all four phases, chosen in random order. The four phases will be: Placebo Phase (microcrystalline cellulose in water), Potassium Chloride Phase (potassium chloride powder in water), Potassium Citrate Phase (potassium citrate powder in water), KMgCit Phase (KMgCit powder in water) During each phase, subjects will receive one of the test drugs for 4 weeks, followed by at least 1 week of withdrawal. Change in 24 hr BP, office BP will be measured at baseline and after each phase. Central aortic blood pressure and carotid-femoral pulse wave velocity, -terminal-telopeptide (CTX), 24 hr urine electrolytes will be measured at 4 weeks in each phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre- or Stage I hypertension, with systolic blood pressure of 120-159 mm and diastolic of 80-99 mm
* Age > 21 years of age

Exclusion Criteria:

* Diabetes mellitus,
* Renal impairment (serum creatinine > 1.4 mg/dL),
* Any heart diseases such as congestive heart failure or sustained arrhythmia,
* Chronic NSAID use,
* Treatment with diuretics,
* Gastroesophageal reflux disease (GERD) requiring treatment with acid reducing agents or antacid more than once a week,
* Esophageal-gastric ulcer,
* Chronic diarrhea
* Hyperkalemia (serum > 4.6 mmol/L for patients on Angiotensin converting enzyme (ACE) inhibitors or Angiotensin receptor blockers (ARB), serum K > 5.0 for patient not on ACE inhibitors or ARBs)
* Liver function test above upper limit of normal range.
* Subjects who require any potassium supplement on a regular basis from any reasons
* Pregnancy
* History of major depression, bipolar disorder, or schizophrenia
* History of substance abuse.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Result] He FJ, Markandu ND, Coltart R, Barron J, MacGregor GA. Effect of short-term supplementation of potassium chloride and potassium citrate on blood pressure in hypertensives. Hypertension. 2005 Apr;45(4):571-4. doi: 10.1161/01.HYP.0000158264.36590.19. Epub 2005 Feb 21. PMID 15723964
- [Result] Conlin PR, Erlinger TP, Bohannon A, Miller ER 3rd, Appel LJ, Svetkey LP, Moore TJ. The DASH diet enhances the blood pressure response to losartan in hypertensive patients. Am J Hypertens. 2003 May;16(5 Pt 1):337-42. doi: 10.1016/s0895-7061(03)00056-6. PMID 12745193
- [Result] He FJ, Marciniak M, Carney C, Markandu ND, Anand V, Fraser WD, Dalton RN, Kaski JC, MacGregor GA. Effects of potassium chloride and potassium bicarbonate on endothelial function, cardiovascular risk factors, and bone turnover in mild hypertensives. Hypertension. 2010 Mar;55(3):681-8. doi: 10.1161/HYPERTENSIONAHA.109.147488. Epub 2010 Jan 18. PMID 20083724
- [Result] Lin PH, Aickin M, Champagne C, Craddick S, Sacks FM, McCarron P, Most-Windhauser MM, Rukenbrod F, Haworth L; Dash-Sodium Collaborative Research Group. Food group sources of nutrients in the dietary patterns of the DASH-Sodium trial. J Am Diet Assoc. 2003 Apr;103(4):488-96. doi: 10.1053/jada.2003.50065. PMID 12669013
- [Result] Lind L, Lithell H, Pollare T, Ljunghall S. Blood pressure response during long-term treatment with magnesium is dependent on magnesium status. A double-blind, placebo-controlled study in essential hypertension and in subjects with high-normal blood pressure. Am J Hypertens. 1991 Aug;4(8):674-9. doi: 10.1093/ajh/4.8.674. PMID 1930849
- [Result] China Salt Substitute Study Collaborative Group. Salt substitution: a low-cost strategy for blood pressure control among rural Chinese. A randomized, controlled trial. J Hypertens. 2007 Oct;25(10):2011-8. doi: 10.1097/HJH.0b013e3282b9714b. PMID 17885542
- [Result] Sellmeyer DE, Schloetter M, Sebastian A. Potassium citrate prevents increased urine calcium excretion and bone resorption induced by a high sodium chloride diet. J Clin Endocrinol Metab. 2002 May;87(5):2008-12. doi: 10.1210/jcem.87.5.8470. PMID 11994333

RESULTS

PARTICIPANT FLOW:
Groups:
- Potassium Magnesium Citrate (KMgCit) Arm: Potassium magnesium citrate will be prepared by mixing potassium citrate, magnesium citrate and/or citric acid by Meta Pharm Development. The content of each sachet will be dissolved in 250 ml water and will be drunk with breakfast and again with dinner during the KMgCit Phase, to deliver 40 meq K, 20 meq Mg and 74 meq citrate per day for 4 weeks
  Potassium magnesium Citrate (KMgCit)
- Potassium Citrate Arm: A special sachet formulation containing 20 meq K/sachet will be made for the study by Meta Pharm Development. The contents of a sachet will be added to 250 ml water and drunk with breakfast and dinner, to deliver 40 meq K (as citrate) per day during the Potassium Citrate Phase for 4 weeks.
  Potassium citrate powder
- Potassium Chloride Arm: Potassium chloride will contain 20 meq KCl per sachet. During the Potassium Chloride Phase, subjects will dissolve the content of each sachet in 250 ml water and ingest it with breakfast and again with dinner, to deliver 40 meq K (as chloride) per day for 4 weeks
  Potassium chloride powder
- Placebo: Placebo will comprise microcrystalline cellulose, equivalent in volume in each sachet as other test products. During the Placebo Phase, subjects will dissolve the entire content of a sachet in 250 ml water and drink it with breakfast and again with dinner for 4 weeks.
  Placebo
Period: KMgCit Phase
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Started | 30 | 0 | 0 | 0
Completed | 30 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: K Citrate Phase
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Started | 0 | 30 | 0 | 0
Completed | 0 | 30 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: KCl Phase
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Started | 0 | 0 | 30 | 0
Completed | 0 | 0 | 30 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Placebo Phase
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Started | 0 | 0 | 0 | 30
Completed | 0 | 0 | 0 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized cross over design so total number of subjects = 30
Groups:
- All Study Participants: Participants took Potassium magnesium Citrate (KMgCit), potassium citrate (KCit), potassium chloride (KCl) and placebo each for 4 weeks in a randomized crossover design.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Average Systolic Blood Pressure
Description: Systolic blood pressure was measured through an ambulatory blood pressure monitoring device worn by each participant for 24 hours after completing each treatment phase. This devise measures blood pressure intermittently throughout the day and night and provides the average of all readings.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 127 (11) | 127 (10) | 126 (9) | 129 (13)

ADVERSE EVENTS:
Arm/Group | Potassium Magnesium Citrate (KMgCit) Arm | Potassium Citrate Arm | Potassium Chloride Arm | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No